CLINICAL TRIAL: NCT05934721
Title: The Mediating Effect of Nociplastic Pain on the Relationship Between Rheumatoid Arthritis Severity and Cognition in Geriatric Patients: A Cross-Sectional Study
Brief Title: Relationship Between Rheumatoid Arthritis Severity and Cognition in the Elderly: The Role of Nociplastic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/282023062023
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis; Rheumatic Diseases; Rheumatoid Polyarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA patients aged 70-90 years: Patients meeting inclusion/exclusion criteria will be recruited from rheumatology clinics and community sources.
  Interventions: Other: Questionnaire and physical assessments

INTERVENTIONS:
Other: Questionnaire and physical assessments — Participants will complete self-report questionnaires assessing pain (CSI) and RA severity (patient global VAS), as well as undergoing physical assessments of RA severity (physician global VAS, swollen/tender joint counts) and cognition (MoCA).

SUMMARY:
this study aims to determine if nociplastic pain mediates the relationship between rheumatoid arthritis (RA) severity and cognitive impairment in geriatric patients 100 patients aged 65-90 years with long-standing RA and assess their disease severity, cognition, and pain sensitization will be recruited. Expectations that patients with more severe RA will have worse cognitive function, and that this relationship will be mediated by higher levels of nociplastic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-90 years
* diagnosed with RA for 10-30 years
* meet ACR/EULAR 2010 criteria

Exclusion Criteria:

* Other inflammatory arthritides
* dementia
* severe depression
* recent corticosteroid or immunosuppressant use

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-dwelling adults aged 65-90 years with a diagnosis of RA for 10-30 years who meet the ACR/EULAR 2010 classification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function as measured by the Montreal Cognitive Assessment (MoCA) | Baseline
  The MoCA assessments cognition in multiple domains; scores ≤26 indicate cognitive impairment. The MoCA is scored out of 30 points, with a higher score indicating better cognitive function. The maximum score on the MoCA is 30, while the minimum score is 0. The test typically takes around 10-15 minutes to complete and is administered by a trained healthcare professional.
Centralized pain as measured by the Central Sensitization Inventory (CSI) | Baseline
  The CSI determines the degree of pain centralization/sensitization. The CSI consists of 25 items that assess various symptoms and experiences associated with CSS, including pain severity and quality, sleep disturbances, fatigue, mood changes, and cognitive difficulties. The CSI is scored on a 0-100 scale, with higher scores indicating a greater degree of central sensitization. A score of 40 or higher is generally considered to indicate the presence of CSS, while a score of 60 or higher indicates a high degree of central sensitization.
RA disease severity as measured by the Physician Global Assessment (0-10 VAS) | Baseline
  Description: 0 = no disease activity; 10 = maximum disease activity

SECONDARY OUTCOMES:
28-joint swollen/tender joint count | Baseline
  Number of joints with swelling/tenderness on examination
Patient Global Assessment (0-10 VAS) | Baseline
  Self-report of RA severity; 0 = no disease activity; 10 = maximum disease activity
Inflammatory markers (ESR) | Baseline
  Markers of inflammation measured through blood tests. ESR is a blood test that measures how quickly red blood cells settle to the bottom of a test tube over a period of one hour. Inflammation in the body can cause red blood cells to clump together, which slows down their settling rate and leads to an elevated ESR. ESR is measured in millimeters per hour (mm/h), and normal values vary depending on age and gender. In general, higher ESR values indicate the presence of inflammation.
Inflammatory markers (CRP) | Baseline
  Markers of inflammation measured through blood tests. CRP is a protein that is produced by the liver in response to inflammation in the body. CRP levels can rise rapidly in response to inflammation, and the test is commonly used to monitor the progression of inflammatory diseases such as rheumatoid arthritis and inflammatory bowel disease. CRP is measured in milligrams per liter (mg/L), and normal values vary depending on age and gender. Higher CRP levels indicate the presence of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No